CLINICAL TRIAL: NCT02199457
Title: An Open Label, Clinical Performance Study to Demonstrate the Clinical Accuracy of the Smartphone Vital Signs System (SVSS)
Brief Title: A Study to Demonstrate the Clinical Accuracy of the Smartphone Vital Signs System (SVSS)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Device development not completed
Sponsor: Léman Micro Devices SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: LMD_CT_001
Record Dates: First submitted 2014-07-11; First posted 2014-07-24 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SVSS and reference devices (Other): Vital signs will be measured on the same subject with the reference devices and with the SVSS. The subject will have blood pressure, pulse, blood oxygen, body temperature and respiration rate measured using standard equipment. The same subject will then use the investigational device which measures all vital signs at the same time, by placing the index finger on a sensor.
  Interventions: Device: SVSS and reference devices

INTERVENTIONS:
Device: SVSS and reference devices — Blood pressure will be measured with standard mercury manometer
Device: SVSS and reference devices — Body temperature taken with infrared thermometer
Device: SVSS and reference devices — Pulse rate and Sp02 measured with a reference pulse oximter. The pulse oximeter is just clipped to the end of the finger.
Device: SVSS and reference devices — Measurement of respiration rate

SUMMARY:
A medical device study to assess the clinical accuracy and equivalence to reference devices of the SVSS to satisfy the requirements of the recognised applicable international standards.

DETAILED DESCRIPTION:
The SVSS is designed to measure and display 5 vital signs: pulse rate, blood oxygen saturation (Sp02), blood pressure, body temperature and respiration rate. These results will be compared for accuracy with the results obtained using standard vital sign measurement equipment on the same subject.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers, male or female, 18 yrs or older, willing and able to participate and sign the informed consent form.

Exclusion Criteria:

* None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-07 (Estimated); Primary Completion 2017-12 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Primary outcome is satisfactory evidence of substantial equivalence of each of the five vital signs with the reference devices within the ranges specified by the standards. | DAY 1
  Accuracy of investigational device compared to the reference devices.

CONTACTS AND LOCATIONS:
Overall Officials: Chris Elliott, Study Director — Sponsor GmbH
Locations (1):
- EPFL, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No